CLINICAL TRIAL: NCT04036552
Title: The Association Between Dietary Choline, Genetics and Anxiety/Depression
Brief Title: The Associations Between Dietary Choline, Genetics and Anxiety/Depression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Other Study IDs: SMEC_2018-19_028
Record Dates: First submitted 2019-03-28; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Choline Deficiency; Anxiety; Depression
MeSH Terms: conditions — Choline Deficiency; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva and blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The associations between dietary choline, genetics and anxiety/depression

DETAILED DESCRIPTION:
Choline, previously considered to be a vitamin, is an essential nutrient involved in a plethora of biological pathways. Choline status is thought to be associated with depression and anxiety, however, the lack of evidence regarding the exact mechanism of its action warrants further investigation. This study aims to explore the associations between dietary choline and depression and anxiety in healthy individuals and how these may differ according to genetics, specifically Phosphatidylethanolamine N-Methyltransferase gene involved in endogenous and exogenous choline metabolism. Establishing these associations could reinforce the need for future intervention trials that could in turn establish causality and determine the mechanistic effects of dietary choline and the PEMT gene activity on depression/anxiety

ELIGIBILITY:
Inclusion Criteria:

* Overall healthy males
* pre-menopausal females of 18-50 years of age.

Exclusion Criteria:

* Individuals with a current clinical diagnosis of anxiety and depression
* pregnant or lactating
* post-menopausal women
* individuals suffering with chronic disease (cardiovascular disease, type-2 diabetes mellitus and cancer)
* individuals using choline, lecithin or soy supplements,
* obese individuals with a Body Mass Index (BMI) >30 kg/m2.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: To be able to detect an association between choline and depression/anxiety required number of participants is 40. However, to reach the adequate balance between groups of people that have the PEMT genetic variant and the ones that do not have it, 80 will be recruited. This is because the PEMT variant of interest is present in 50% of the population
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-10-03 (Estimated); Study Completion 2019-10-03 (Estimated)

PRIMARY OUTCOMES:
Depression | 1 day observation
  Hospital Anxiety and Depression questionnaire score higher than 11
Anxiety | 1 day observation
  Hospital Anxiety and Depression questionnaire score higher than 11

SECONDARY OUTCOMES:
Choline intake | 3 day observation
  Dietary choline intake
Plasma choline levels | 1 measurement
  Choline levels in plasma obtained by colorimetry

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's University, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No